CLINICAL TRIAL: NCT05753397
Title: The Intertransverse Process Block - Single or Multiple Injection? A Randomised, Procedure Related, Blinded Crossover Trial in Healthy Volunteers
Brief Title: ITP Block: Single or Multiple Injection?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZUH-ITP-MBCS
Record Dates: First submitted 2023-02-08; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia, Local
Keywords: ultrasound guided nerveblock; Intertransverse Process Block; Healthy volunteers; Thoracic dermatomes; sensory mapping
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single injection (Experimental): 1x21ml Ropivacaine (7.5mg/ml) at ITTC T4. Including two sham injections at ITTC T2 and ITTC T6
  Interventions: Drug: Ropivacaine injection
- Multiple injection (Experimental): 3x7ml Ropivacaine (7.5mg/ml) at ITTC T2, T4 and T6.
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — We are testing if single injection Ropivacaine is non-inferior to multiple-injection Ropivacaine when applied within the intertransverse tissue complex (that is: a paraspinal application mimicking the paravertebral block)

SUMMARY:
The intertransverse process (ITP) block is a new ultrasound-guided peripheral nerve block modality designed for peri- and postoperative pain amelioration for patients undergoing surgery on the thoracic wall. The modality mimics the well-known thoracic paravertebral block but, potentially, with a significantly lower risk of adverse events. However, evidence for the ITP block efficacy and the clinical applicability, e.g. the number of injections, dermatomal coverage etc., is still sparse and needs further investigation.

In this noninferiority, short-term, randomised, blinded, procedure-related crossover trial we will further investigate the ITP block in healthy volunteers to see whether it is possible to reduce the number of injections from three to one and substantiate the number of anaesthetised dermatomes with either modality as the primary outcome. Secondary outcomes include sensory mapping of the thorax, non-invasive thermography, changes in non-invasive blood pressure and satisfaction with block application.

At Zealand University Hospital, twelve healthy volunteers will be randomised to receive either a single injection or multiple injection blockade with long-lasting local anaesthetic. All twelve participants will, on day one, receive active blockade with the well-known marketed drug Ropivacaine 7.5mg/ml, and all participants will receive 21 ml; that is six participants receiving 1x21ml and six participants receiving 3x7ml. The six participants receiving 1x21 ml will also receive two sham injections to ensure the blinding. No placebo is used. On day two the intervention is crossed over and the participants will receive the other modality. Within the following hour after block application, relevant standard cutaneous testing is performed; pinprick and cold sensation test for dermatomal coverage, the anaesthetised skin area is pen marked on the thorax and photo documented, thermography to measure temperature differences between each hemi thorax (blocked side vs. non- blocked side) and standard non-invasive blood pressure measurements are performed.

After 60 minutes of relevant testing the trial ends and the participant are free to leave the hospital 2 hours after block application if no adverse events are recorded. With such series of test procedures, we will generate new knowledge of the ITP block before future patients undergo breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

Male sex Age ≥ 18 years at the date of inclusion American Associations of Anaesthesiologist (ASA) class I-II Have received thorough information, orally and in written form, and signed the "Informed Consent" form on participation in the study.

Weight > 52,5 kilograms (chosen due to the international maximal single dose of Ropivacaine (3mg/kg))

Exclusion Criteria:

* Substantial co-morbidity: American Associations of Anaesthesiologist (ASA) class > II
* Inability to speak and understand Danish
* Inability to cooperate
* Allergy to study drugs
* Daily intake of analgesics (investigators decision)
* Alcohol and/or drug overuse (investigators decision)
* Previous thoracic trauma or thoracic surgery
* Previous/current piercing of the nipple of any kind on blockade side
* Tattoos on the thorax (according to the investigators decision)
* Any systemic muscular or neuromuscular disease
* Any use of vasodilatory substance (investigators decision)
* Local infection at the site of injection or systemic infection
* Difficult sonoanatomical visualisation of the target area (SCTL, ITTC etc.) necessary for the block execution
* Severe hypovolemia

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-26 (Estimated); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Anesthetized thoracic dermatomes. | Minute 35 post block application.
  The primary outcome of this procedure related study is the number of anesthetized thoracic dermatomes.
  Key points of sensory testing will follow International Standards for Neurological Classification of Spinal Cord Injury.
  Dermatomal spread of the single- and multiple-injection ITP blocks will be determined using both mechanical (pinprick) and temperature (cold) discrimination, deficit for either modality is regarded as a sensory deficit.

SECONDARY OUTCOMES:
Sensory mapping. | Minute 45 post block application.
  The extent of cutaneous spread of the sensory block (single vs multiple-injection ITP block). Spread of the single- and multiple-injection ITP blocks respectively will be determined using both mechanical (pinprick) and temperature (cold) discrimination, deficit for either modality is regarded as a sensory deficit. Relevant areas are marked on the participants' thoraxes and transferred to paper for conversion to square centimeters.
Thermography in a clinical setup. | Minutes 10, 20 and 30 post block application
  A peripheral nerve block leads to a motor and somatosensory blockade but also sympathetic nerve fibers are being blocked. The following sympatholysis increases the diameter of the vessels (vasodilatation) in the skin and thereby increasing the blood flow and increases the temperature. Hence, it is possible that the technique would help determine the expected success of the blockade in a fast and efficient manner.
  We will use the "Testo 883 Thermography camera" (Testo SE & Co. KGaA, Lenzkirch, Baden-Württemberg, Germany) to obtain infrared imaging of the anterior thorax of the participants. Each thoracic dermatome from T2-T10 will be evaluated in the mid-clavicular line and reported as the temperature difference when compared to the contralateral side.
Non-invasive blood pressure. | Minutes 15, 30 and 60 post block application.
  Standard non-invasive blood pressure measurement reported as mean arterial pressure.
Block application satisfaction. | During block application.
  The Numeric Rating Scale (NRS) for pain scores is a well-known clinical scale. It ranges 0-10, 0 being no pain and 10 being the worst pain imaginable.
  The participant will rate the block application NRS score orally during block application.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Zealand University Hospital, Roskilde, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No